CLINICAL TRIAL: NCT02980237
Title: Effectiveness of an e-Health Program at Workplace in the Promotion of Quality of Life of Office Workers: Protocol of a Randomized Controlled Trial by Cluster
Brief Title: e-Health Education Program at Workplace
Acronym: e-Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rosimeire Simprini Padula (Other)
Responsible Party: Sponsor-Investigator, Rosimeire Simprini Padula, PhD, Universidade Cidade de Sao Paulo
Organization: Universidade Cidade de Sao Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1.023.328
Record Dates: First submitted 2016-08-23; First posted 2016-12-02 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Health Behavior
Keywords: Office workers; Quality of life; e-Learning; Occupational health
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eHealth_additional support (Experimental): An e-learning education program whose audiovisual content will be implemented. The course could be access in the workplace but they will be additional support.
  Interventions: Other: eHealth_additional support
- eHealth (Active Comparator): This group will receive an e-learning education program same as the intervention group . However, the participants will not receive additional support by team.
  Interventions: Other: eHealth_program

INTERVENTIONS:
Other: eHealth_additional support — An e-learning education program whose audiovisual content will be implemented. Nine audiovisual e-Health program will be composed of nine video classes addressing the following topics: 1) musculoskeletal health, 2) healthy diet and 3) mental health were identified through focus group. A communication tool will be adopted is the Moodle environment. All the participants will be able to whipping the web platform and questions regarding access and navigation are answered by e-mail. All participants will be monitored, as viewing the videos, and whenever it is identified that the participants not accessed and lack of interest of reasons. A team of tutors will be responsible for online support providing reinforcing stimuli and clarifying any questions (intervention group) on the content.
  Arms: eHealth_additional support
Other: eHealth_program — The comparative group will receive the same eHealth education program that intervention group. But the comparative group will receive only audiovisuals without additional support. .
  Arms: eHealth

SUMMARY:
The objective this study is evaluate if an e-Health education program at the workplace to contributes to improve quality of life from Office Workers. And:Life style modification; Improve physical activity Reduces on Anthropometric Measures; Reduces Pain and discomfort in the musculoskeletal system

DETAILED DESCRIPTION:
Objective: The purpose of this study is evaluate the effectiveness of an e-Health education program at the workplace in the quality of life promotion.

Design: Double Blinded. Randomized clinical trial by cluster. Setting: Office Workers of the Universidade Publica do Estado da Bahia, Bahia State, Brazil. Participants: 348 office workers are enrollment, both sex, with over 18 year old.

Intervention: Participants will randomized in: (1) reference group will receive an e-learning health education compose by nine video-class according to the dimensions: 1) musculoskeletal health, 2) eating health e 3) mental health. A video will available by moodle platform every 20 days during six months. In this period the workers will monitored regarding to access the videos and and reinforcements to remain in the program. (2) intervention group: they will receive e-health education program with additional support healthcare tutor everyday.

ELIGIBILITY:
Inclusion Criteria:

* Technical-administrative workers, computer users for a minimum period of six months. ,
* Signed informed consent form

Exclusion Criteria:

* Suspected or confirmed pregnant workers at randomization time
* Mothers what Breastfeeding
* Workers in annual leave.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2017-10-17 (Actual); Study Completion 2018-03-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline Quality of life at 6 and 8 months | Baseline, 6 and 8 months
  A questionnaire to evaluate the improve the quality of life after 6 and 8 months after began the program will be used (WHOQOL-BREF :instrument comprises 26 items, which measure the following broad domains: physical health, psychological health, social relationships, and environment).

SECONDARY OUTCOMES:
Change from Anthropometric measure at 6 and 8 months | Baseline, 6 and 8 months
  Changes on anthropometric measurements (weight, abdominal circumference, waist circumference, hip circumference, body mass and height). For this study, body mass index (BMI), body fat percentage (BFP) and waist-hip ratio will be used and assessment 6 and 8 months after starting the eHealth program.
Change from Pain and/or musculoskeletal discomfort measure at 6 and 8 months | Baseline, 6 and 8 months
  To assessement the intensity of musculoskeletal complains (pain and discomfort) in baseline and 6 and 8 months an after starting the eHealth program.
Change from Lifestyle at 6 and 8 months | Baseline, 6 and 8 months
  Change in health behavior, in physical activity level (min/week) after starting the eHealth program in 6 and 8 months will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Rosimeire S Padula, PhD, Study Director — Universidade Cidade de São Paulo
Locations (1):
- Rosimeire Simprini Padula, Atibaia, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Andersen JH, Fallentin N, Thomsen JF, Mikkelsen S. Risk factors for neck and upper extremity disorders among computers users and the effect of interventions: an overview of systematic reviews. PLoS One. 2011 May 12;6(5):e19691. doi: 10.1371/journal.pone.0019691. PMID 21589875
- [Result] Dillon C, Petersen M, Tanaka S. Self-reported hand and wrist arthritis and occupation: data from the U.S. National Health Interview Survey-Occupational Health Supplement. Am J Ind Med. 2002 Oct;42(4):318-27. doi: 10.1002/ajim.10117. PMID 12271479
- [Result] Mulder R, Pouwelse M, Lodewijkx H, Bolman C. Workplace mobbing and bystanders' helping behaviour towards victims: the role of gender, perceived responsibility and anticipated stigma by association. Int J Psychol. 2014 Aug;49(4):304-12. doi: 10.1002/ijop.12018. Epub 2013 Nov 20. PMID 24990642
- [Result] Raman SR, Al-Halabi B, Hamdan E, Landry MD. Prevalence and risk factors associated with self-reported carpal tunnel syndrome (CTS) among office workers in Kuwait. BMC Res Notes. 2012 Jun 13;5:289. doi: 10.1186/1756-0500-5-289. PMID 22695029
- [Result] Thorp AA, Owen N, Neuhaus M, Dunstan DW. Sedentary behaviors and subsequent health outcomes in adults a systematic review of longitudinal studies, 1996-2011. Am J Prev Med. 2011 Aug;41(2):207-15. doi: 10.1016/j.amepre.2011.05.004. PMID 21767729
- [Result] Waersted M, Hanvold TN, Veiersted KB. Computer work and musculoskeletal disorders of the neck and upper extremity: a systematic review. BMC Musculoskelet Disord. 2010 Apr 29;11:79. doi: 10.1186/1471-2474-11-79. PMID 20429925
- [Result] Bernal D, Campos-Serna J, Tobias A, Vargas-Prada S, Benavides FG, Serra C. Work-related psychosocial risk factors and musculoskeletal disorders in hospital nurses and nursing aides: a systematic review and meta-analysis. Int J Nurs Stud. 2015 Feb;52(2):635-48. doi: 10.1016/j.ijnurstu.2014.11.003. Epub 2014 Nov 15. PMID 25480459
- [Result] Bandoni DH, Sarno F, Jaime PC. Impact of an intervention on the availability and consumption of fruits and vegetables in the workplace. Public Health Nutr. 2011 Jun;14(6):975-81. doi: 10.1017/S1368980010003460. Epub 2010 Dec 21. PMID 21205408
- [Result] Cash SW, Beresford SA, Henderson JA, McTiernan A, Xiao L, Wang CY, Patrick DL. Dietary and physical activity behaviours related to obesity-specific quality of life and work productivity: baseline results from a worksite trial. Br J Nutr. 2012 Sep 28;108(6):1134-42. doi: 10.1017/S0007114511006258. Epub 2011 Dec 6. PMID 22142517
- [Result] Knies S, Boonen A, Severens JL. Do the Washington Panel recommendations hold for Europe: investigating the relation between quality of life versus work-status, absenteeism and presenteeism. Cost Eff Resour Alloc. 2014 Nov 24;12:24. doi: 10.1186/1478-7547-12-24. eCollection 2014. PMID 25904824
- [Result] Robroek SJ, Polinder S, Bredt FJ, Burdorf A. Cost-effectiveness of a long-term Internet-delivered worksite health promotion programme on physical activity and nutrition: a cluster randomized controlled trial. Health Educ Res. 2012 Jun;27(3):399-410. doi: 10.1093/her/cys015. Epub 2012 Feb 20. PMID 22350194
- [Result] Kreps GL, Neuhauser L. New directions in eHealth communication: opportunities and challenges. Patient Educ Couns. 2010 Mar;78(3):329-36. doi: 10.1016/j.pec.2010.01.013. Epub 2010 Mar 3. PMID 20202779
- [Result] Tate DF, Jackvony EH, Wing RR. A randomized trial comparing human e-mail counseling, computer-automated tailored counseling, and no counseling in an Internet weight loss program. Arch Intern Med. 2006 Aug 14-28;166(15):1620-5. doi: 10.1001/archinte.166.15.1620. PMID 16908795
- [Result] Palmer KT, Harris EC, Linaker C, Barker M, Lawrence W, Cooper C, Coggon D. Effectiveness of community- and workplace-based interventions to manage musculoskeletal-related sickness absence and job loss: a systematic review. Rheumatology (Oxford). 2012 Feb;51(2):230-42. doi: 10.1093/rheumatology/ker086. Epub 2011 Mar 16. PMID 21415023
- [Result] Krukowski RA, Tilford JM, Harvey-Berino J, West DS. Comparing behavioral weight loss modalities: incremental cost-effectiveness of an internet-based versus an in-person condition. Obesity (Silver Spring). 2011 Aug;19(8):1629-35. doi: 10.1038/oby.2010.341. Epub 2011 Jan 20. PMID 21253001
- [Result] Bennell KL, Rini C, Keefe F, French S, Nelligan R, Kasza J, Forbes A, Dobson F, Abbott JH, Dalwood A, Vicenzino B, Harris A, Hinman RS. Effects of Adding an Internet-Based Pain Coping Skills Training Protocol to a Standardized Education and Exercise Program for People With Persistent Hip Pain (HOPE Trial): Randomized Controlled Trial Protocol. Phys Ther. 2015 Oct;95(10):1408-22. doi: 10.2522/ptj.20150119. Epub 2015 May 28. PMID 26023213
- [Derived] Tosta Maciel RRB, Chiavegato LD, Camelier FW, Portella DD, De Souza MC, Padula RS. Does tutors' support contribute to a telehealth program that aims to promote the quality of life of office workers? A cluster randomized controlled trial. Contemp Clin Trials Commun. 2021 Feb 1;21:100722. doi: 10.1016/j.conctc.2021.100722. eCollection 2021 Mar. PMID 33604486